CLINICAL TRIAL: NCT06438484
Title: The Challenges of Evidence-based Prehabilitation in a Real-life Context for Patients Preparing for Colorectal Surgery - a Cohort Study and Multiple Case Analysis
Brief Title: The Challenges of Evidence-based Prehabilitation in a Real-life Context for Patients Preparing for Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, Aletta Danielle Talen, Mac clinical health scientist, Nij Smellinghe Hosptial
Other Study IDs: NUTNS
Record Dates: First submitted 2024-05-15; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Surgery
Keywords: Preoperative Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low risk: Patients with high aerobic capacity and good nutritional status were given the advice to eat healthy and stay active until surgery. Postoperative data were collected for evaluative purposes.
- High risk: High-risk patients followed an evidence-based multimodal prehabilitation program for five weeks, incorporating modalities tailored to address their impairments. Patients performed physical exercise training and/or received dietary counseling for five weeks, provided by a trained physiotherapist and dietitian (both >15 years experience).
  Interventions: Behavioral: multimodal prehabilitation program

INTERVENTIONS:
Behavioral: multimodal prehabilitation program — Patients performed physical exercise training and/or received dietary counseling for five weeks, provided by a trained physiotherapist and dietitian (both >15 years experience). The physical exercise training consisted of high-intensity interval training (HIIT) three times a week and functional strengthening exercises. Patients visited the hospital two times a week and performed home exercise training five times a week on a stationary cycle ergometer (Corival Home+, Lode BV, Groningen, The Netherlands).
  The dietary intervention consisted of optimization of energy and protein intake, optimization of timing of eating protein-rich products, and if necessary additional protein and vitamin supplements. Individual protein requirements were set at 1.5-1.9 g/kg fat free mass. Patients used the eiFIT-application or a food diary to track their protein intake.
  Groups: High risk

SUMMARY:
Background: Multimodal prehabilitation programs are effective in reducing complications after colorectal surgery in patients with high risk of postoperative complications due to low aerobic capacity and/or malnutrition. However, high implementation fidelity is needed to achieve these effects in real-life practice. Therefore, this study aimed to investigate the implementation fidelity of an evidence-based prehabilitation program in the real-life context of a regional hospital.

Methods: In this observational cohort study with multiple case analysis, we enrolled all patients who underwent surgery for colorectal cancer from January 2023 to June 2023, in one Dutch peripheral hospital. Patients meeting criteria for low aerobic capacity or malnutrition were advised to participate in a personalized prehabilitation program. Implementation fidelity was investigated on four domains; 1) coverage (participation rate), 2) duration (number of days following the prehabilitation program), 3) content (delivery of prescribed intervention modalities), and 4) frequency (attendance of sessions and compliance with prescribed parameters). An aggregated percentage of content and frequency was calculated to determine overall adherence. The intended outcomes were improvement in preoperative aerobic capacity and malnutrition, and improved postoperative recovery (i.e., reducing complications, length of stay, and time to functional recovery).

DETAILED DESCRIPTION:
Study design and patients This observational cohort study was conducted from January 2023 to June 2023 with case analysis on the high-risk patients following the prehabilitation program in Nij Smellinghe (NS). The study was approved by the Local Ethic Committee of NS. The first author was a physiotherapist, who acted as an embedded scientist in the colorectal pathway25. For the period of this study, only one physiotherapist and dietitian performed the prehabilitation program to prevent provider-dependent bias. All patients, both high-risk and low-risk, of 18 years or older scheduled for elective colorectal surgery in NS were asked for their informed consent to be included in the cohort. No exclusion criteria were applied. The STrengthening the Reporting of Observational Studies in Epidemiology (STROBE) guideline for reporting observational studies was followed26.

Study setting NS is a regional hospital with 339 beds in The Netherlands, where annually 150 patients undergo colorectal surgery27. NS is an innovative hospital in the field of perioperative care and the Enhanced Recovery After Surgery (ERAS) protocol has been implemented into usual care since 201828. In January 2023, following new scientific insights, an evidence-based multimodal prehabilitation program was implemented in the colorectal pathway. This pathway included assessment of patients on their risk of postoperative complications and offering a multimodal prehabilitation program for high-risk patients.

Preoperative risk assessment When patients were indicated for colorectal surgery, a physiotherapist and dietitian conducted risk assessment for postoperative complications. Patients meeting criteria for low aerobic capacity and/or high risk of malnutrition were advised to participate in a personalized prehabilitation program2,29.

The physiotherapist assessed aerobic capacity. Aerobic capacity was measured by the cardiopulmonary exercise test (CPET) or modified steep ramp test (SRT), following the protocol of previous research on preoperative risk assessment2,15,30. Patients with a low aerobic capacity, indicated by a work at peak exercise achieved at the modified SRT ≤1.5W/kg or an oxygen uptake at the VAT ≤11mL/kg/min at the CPET, were indicated as high-risk patients.

The dietitian evaluated risk of malnutrition by using the Patient-Generated Subjective Global Assessment Short Form (PG-SGA SF). Based on the Global Leadership Initiative on Malnutrition (GLIM) criteria, patients were diagnosed with malnutrition, thus indicating the nutrition-modality of prehabilitation31. According to the GLIM-criteria, malnutrition is defined as the presence of one phenotypic criterion (non-volitional weight loss, low body mass index, and reduced muscle mass) and one etiologic criterion (reduced food intake or assimilation, and inflammation or disease burden)32. Muscle mass and body composition was assessed with the bioelectrical impedance analysis (BIA) (Bodygram Plus, Akern, Italy).

Patients with high-risk profile: multimodal prehabilitation program High-risk patients followed an evidence-based multimodal prehabilitation program for five weeks, incorporating modalities tailored to address their impairments2,12,15. Patients performed physical exercise training and/or received dietary counseling for five weeks, provided by a trained physiotherapist and dietitian (both >15 years experience). The physical exercise training consisted of high-intensity interval training (HIIT) three times a week and functional strengthening exercises. Patients visited the hospital two times a week and performed home exercise training five times a week on a stationary cycle ergometer (Corival Home+, Lode BV, Groningen, The Netherlands).

The dietary intervention consisted of optimization of energy and protein intake, optimization of timing of eating protein-rich products, and if necessary additional protein and vitamin supplements. Individual protein requirements were set at 1.5-1.9 g/kg fat free mass. Patients used the eiFIT-application or a food diary to track their protein intake33.

Treating patients with low hemoglobin levels, offering alcohol- and smoking cessation interventions, and giving psychological support were also elements of the prehabilitation program in NS. However, this is already part of usual care since implementation of the ERAS-protocol and therefore not specifically evaluated in this study. A detailed description of the complete pathway is provided in Appendix 1.

Statistical analysis All data were analyzed using descriptive statistics. For patient characteristics continuous data were tested for normality by the Shapiro-Wilk test and QQ-plot. Median and interquartile range (IQR) or mean and standard deviation were reported accordingly. To report the fidelity of the prehabilitation program, absolute values and percentages were given. To prevent selection bias, NS reimbursed the expenses of prehabilitation for people who otherwise could not afford it, as insurance companies did not reimburse prehabilitation in The Netherlands during the study period. Data were analyzed using R Framework 4.2.2 for macOS (version 2022, Vienna)42.

ELIGIBILITY:
Inclusion Criteria:

* a patient must be awaiting CRC surgery in NS
* be 18 years or older

Exclusion Criteria:

* Patient data will only be excluded if they do not permit the usage of their data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients following the prehabilitation program in Nij Smellinghe
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Coverage | january 2023 - june 2023
  Coverage was defined as 'the participation rate in the innovation by the intended audience' and was determined as the percentage of eligible patients who were assessed and able to follow the suitable prehabilitation pathway. Reasons for drop-out and non-participation were reported.
Duration | january 2023 - june 2023
  , which can be subdivided into coverage, duration, content, and frequency. Duration was measured by the number of days between assessment and surgery and should be at least thirty days.
Content | january 2023 - june 2023
  Content was measured by the number of different components of the intervention delivered.
Frequency | january 2023 - june 2023
  Frequency was measured by the percentage of times when the training intensity as prescribed, time, and the days on which nutritional requirements were achieved

SECONDARY OUTCOMES:
Preoperative aerobic capacity | january 2023 - june 2023
  Preoperative aerobic capacity was measured before and after the prehabilitation program by the Steep Ramp Test. The maximum wattage will be reported.
Preoperative nutritional status | january 2023 - june 2023
  Preoperative risk of malnutrition was measured before and after the prehabilitation program by the the patient generated subjective global assessment short form (PG-SGA SF). This is a validated instrument used by dietitians for the assessment of malnutrition and monitoring of interventions. A low score means a low risk of malnutrition.
Complications | january 2023 - june 2023
  The occurrence of complications was reported, and complications were categorized according to the Clavien-Dindo classification.
Length of stay | january 2023 - june 2023
  Length of stay was defined as days admitted to the hospital2.
Time to recovery of physical functioning | january 2023 - june 2023
  Time to recovery of physical functioning was measured by the modified Iowa level of assistance scale (mILAS) and was reported as time in days between surgery and full inhospital recovery of physical functioning.
Facilitation strategies | january 2023 - june 2023
  Facilitation strategies are strategies to optimize implementation aimed at barriers known from previous research, which are logistical and financial challenges. The physiotherapist, dietitian and embedded researcher documented their observations on influencing factors in a logbook.
Practitioner responsiveness | january 2023 - june 2023
  Practitioner responsiveness is defined as 'engagement to the intervention'. Practitioner responsiveness was measured by a short questionnaire for the physiotherapist and dietitian based on a measurement instrument for determinants of innovation at the end of the study period. Participant responsiveness was measured by a short questionnaire after finishing their prehabilitation program, based on questionnaires in comparable studies
Participant responsiveness | january 2023 - june 2023
  Participant responsiveness is defined as 'engagement to the intervention'. Participant responsiveness was measured by a short questionnaire after finishing their prehabilitation program, based on questionnaires in comparable studies

OTHER OUTCOMES:
patiënt characteristics, age | january 2023 - june 2023
  age(years)
patiënt characteristics, sex | january 2023 - june 2023
  sex (male or female)
patiënt characteristics, living situation | january 2023 - june 2023
  living situation(together or alone)
patiënt characteristics, BMI | january 2023 - june 2023
  body mass index(BMI)
patiënt characteristics, comorbidities | january 2023 - june 2023
  comorbidities(age-adjusted Charlson Comorbidity index)
patiënt characteristics, hb | january 2023 - june 2023
  haemoglobin level(mmol/L)
patiënt characteristics, tumor location | january 2023 - june 2023
  tumor location(rectal or colon)
patiënt characteristics, ASA | january 2023 - june 2023
  ASA score(I-IV)
patiënt characteristics, surgical procedure | january 2023 - june 2023
  surgical procedure (open or laparoscopic)

CONTACTS AND LOCATIONS:
Overall Officials: Aletta Danielle Talen, drs, Principal Investigator — Nij Smellinghe
Locations (1):
- Nij Smellinghe hospital, Drachten, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data are pseudonymized and stored in a secured environment. The data that support the findings of this study are available from Nij Smellinghe, but restrictions apply to the availability of these data, which were used under license for the current study, and so are not publicly available. Data are however available from the authors upon reasonable request and with permission of Nij Smellinghe.

REFERENCES:
- [Derived] Talen AD, van Meeteren NLU, Barten JA, Pereboom I, Krijnen WP, Jager-Wittenaar H, Bongers BC, van der Sluis G. The challenges of evidence-based prehabilitation in a real-life context for patients preparing for colorectal surgery-a cohort study and multiple case analysis. Perioper Med (Lond). 2025 Jan 17;14(1):7. doi: 10.1186/s13741-024-00481-w. PMID 39825452